CLINICAL TRIAL: NCT06992193
Title: Is Digital Anesthesia a Viable Alternative for Pain and Anxiety Control in Paediatric Dentistry?
Brief Title: Effectiveness of Digital Anesthesia Versus Conventional Techniques in Reducing Pain and Anxiety in Children
Acronym: DAPAED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Alp Abidin Ateşçi, DDS, PhD, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alp; 24-11/83 (Other Grant/Funding Number: Ethics Committee on Human Research, Ege University)
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pain in Pediatric Dentistry; Dental Anxiety
Keywords: Dental Anxiety; Pain Management; Intraosseous anesthesia; Local Anesthesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Digital Anesthesia (Experimental): Children receiving intraosseous local anesthesia via a computer-controlled delivery system (SleeperOne 5®) using 4% articaine with 1:200,000 epinephrine.
  Interventions: Device: Digital Anesthesia
- Infiltration Anesthesia (Active Comparator): Children receiving traditional infiltration anesthesia using 2% lidocaine with 1:100,000 epinephrine via standard dental syringe.
  Interventions: Drug: Infiltration Anesthesia
- Mandibular Block Anesthesia (Active Comparator): Children receiving conventional inferior alveolar nerve block with 2% lidocaine and 1:100,000 epinephrine using a long dental needle.
  Interventions: Drug: Mandibular Block

INTERVENTIONS:
Device: Digital Anesthesia — Computer-controlled intraosseous anesthesia system (Dental Hi Tec, France) used to deliver 1.3 mL of 4% articaine with 1:200,000 epinephrine in two stages: gingival and intraosseous injection. The system provides consistent flow and reduced pain perception in children.
  Other Names: SleeperOne 5
  Arms: Digital Anesthesia
Drug: Infiltration Anesthesia — 1 mL of 2% lidocaine with epinephrine was delivered via buccal infiltration using a conventional aspirating syringe and 27-gauge short needle. Topical benzocaine gel was applied for 30 seconds prior to injection.
  Other Names: Lidocaine hydrochloride 2% with epinephrine 1:100,000
  Arms: Infiltration Anesthesia
Drug: Mandibular Block — 1 mL of lidocaine was administered using the inferior alveolar nerve block technique via a conventional dental syringe and 27-gauge long needle. Negative aspiration was confirmed prior to slow deposition.
  Other Names: IANB
  Arms: Mandibular Block Anesthesia

SUMMARY:
This multicenter randomized controlled clinical trial was conducted to evaluate the effectiveness of digital anesthesia using a computer-controlled intraosseous system (SleeperOne 5®) compared to traditional local anesthesia techniques (infiltration and mandibular block) in paediatric dental patients.

A total of 79 children aged 6-12 years were randomly assigned to one of three groups. Pain perception, anxiety levels, and behavioral responses were assessed using validated tools including the Wong-Baker FACES Pain Scale, the Modified Child Dental Anxiety Scale (MCDAS), and the FLACC behavioral scale.

The study aimed to determine whether digital anesthesia could provide a less painful and less anxiety-inducing experience for children during dental treatment. Findings may support broader clinical adoption of computer-assisted anesthetic delivery in paediatric dentistry.

DETAILED DESCRIPTION:
This randomized controlled clinical trial was designed to compare the effects of digital anesthesia, conventional infiltration, and mandibular block techniques on pain perception, anxiety levels, and behavioral responses in paediatric dental patients. The study was conducted at two academic institutions: Ege University and Beykent University in Turkey.

A total of 79 healthy, cooperative children aged 6 to 12 years requiring restorative, endodontic, or extraction procedures on primary teeth were randomly assigned to one of three anesthesia groups: digital anesthesia (n=34), infiltration (n=22), and mandibular block (n=23). Randomization was performed using a computer-generated sequence, and pain, anxiety, and behavior were assessed by a blinded, calibrated examiner.

The digital anesthesia group received intraosseous injection via the SleeperOne 5® system (using 4% articaine with 1:200,000 epinephrine). The infiltration and block groups received 2% lidocaine with 1:100,000 epinephrine using conventional syringes. All patients received topical 20% benzocaine gel prior to injection.

Pain was assessed at three time points (needle insertion, anesthetic delivery, and treatment) using the Wong-Baker FACES scale. Dental anxiety was measured pre- and post-treatment using the Modified Child Dental Anxiety Scale (MCDAS), and behavioral responses were recorded during treatment using the FLACC scale.

The aim was to evaluate whether digital anesthesia provides superior outcomes in terms of comfort, reduced fear, and improved cooperation in the paediatric dental setting.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years
* ASA I or II health status
* Cooperative behavior (Frankl score 3-4 or Venham score 0-2)
* Indicated for restorative, endodontic, or extraction treatment on primary teeth
* No prior local anesthesia experience during the previous 6 months

Exclusion Criteria:

* Presence of systemic or neurological diseases
* Use of analgesics within 48 hours before the procedure
* Uncooperative behavior (Frankl score 1-2 or Venham score >2)
* Incomplete cooperation during the procedure
* Allergy to articaine, lidocaine, or epinephrine

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES pain scores at three time points | Time Frame: Immediately before needle insertion, during anesthetic delivery at the time of the procedure, and during dental procedure (Day 1)
  Pain was assessed using the Wong-Baker FACES Pain Rating Scale at three stages: (1) needle insertion, (2) anesthetic delivery, and (3) during dental treatment. Scores range from 0 (no hurt) to 10 (hurts worst).

SECONDARY OUTCOMES:
Change in MCDAS anxiety scores before and after treatment | Day 1 - immediately before and after dental procedure
  Dental anxiety was measured using the Modified Child Dental Anxiety Scale (MCDAS) immediately before and after the procedure. The scale ranges from 8 to 40, with higher scores indicating greater anxiety.
FLACC behavioral pain scores during anesthesia | Periprocedural (Day 1) - during anesthetic injection phase
  Behavioral responses were recorded using the FLACC scale, which evaluates Face, Legs, Activity, Cry, and Consolability. Each domain is scored from 0-2, for a total range of 0-10.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Beykent University Faculty of Dentistry Department of Pediatric Dentistry, Istanbul
  - Ege University Faculty of Dentistry Department of Pediatric Dentistry, Izmir

REFERENCES:
- [Derived] Atesci AA, Korkut Isik B, Yilmaz DO, Gergit B, Kilic MC, Oncag RO. Is Digital Anesthesia a Viable Alternative for Pain and Anxiety Control in Pediatric Dentistry? Int J Paediatr Dent. 2025 Oct 25. doi: 10.1111/ipd.70048. Online ahead of print. PMID 41137566